CLINICAL TRIAL: NCT02399358
Title: Factors Associated With Hyponatremia Induced by High-dose Cyclophosphamide: Prospective Cohort Study
Brief Title: Factors Associated With Hyponatremia Induced by High-dose Cyclophosphamide
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Diego Hernan Giunta, MD (Other)
Responsible Party: Sponsor-Investigator, Diego Hernan Giunta, MD, Investigator, Hospital Italiano de Buenos Aires
Organization: Hospital Italiano de Buenos Aires (Other)
Other Study IDs: 2439
Record Dates: First submitted 2015-03-22; First posted 2015-03-26 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Hyponatremia
Keywords: Drug induced Hyponatremia; Cyclophosphamide; Hyponatremia; Cyclophosphamide induced Hyponatremia
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- High-dose Cyclophosphamide: Patients requiring infusion of high-dose cyclophosphamide in the period 2015-2017 will be included. After informed consent, patients will de follow up from the infusion of cyclophosphamide to 30 days after hospital discharge.

SUMMARY:
Prospoctive cohort of high-dose cyclophosphamide exposed patients. With active estandardize screening of hyponatremia development in the follow up period.

DETAILED DESCRIPTION:
Primary objectives

1. To identify the factors associated with the development of hyponatremia in patients receiving high-dose cyclophosphamide (2.5 grams or more).
2. Generate and validate a predictive score of developing hyponatremia high-dose cyclophosphamide.
3. To estimate the incidence of hyponatremia in patients undergoing high-dose cyclophosphamide.

Study design. Observational prospective cohort study of Patients after infusion of high-dose cyclophosphamide. Follow up period will be from cyclophosphamide infusion until one month after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over 18 years) who were admitted to the Hematology / Oncology and Medical Clinic Hospital Italiano de Buenos Aires infusion of high-dose cyclophosphamide for conducting MSCH prior BMT, GATLA and HyperCVAD in the period 2015-2017.

Exclusion Criteria:

* Refusal to participate or to the process of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (Over 18 years) admitted for high-dose cyclophosphamide.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Hyponatremia | Between 6 and 8 hours after the infusion of cyclophosphamide is performed.
  Hyponatremia, measured as any value sodium after infusion and defined as positive if sodium less than 135 mEq / l (Yes / No, dichotomous categorical variable). For the incidence of hyponatremia is only included in the calculation hionatremia patients with normal sodium before infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Warley, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Belen Bonella, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Victoria Otero, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Bruno L Ferreyro, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Peron 4190, Buenos Aires, Buenos Aires F.D., Argentina